CLINICAL TRIAL: NCT04568694
Title: Planned Semi-Elective Lung Transplantation Using 10C Cold Static Preservation: A Proof-of-Concept Study
Brief Title: Planned Semi-Elective Lung Transplantation Using 10C Cold Static Preservation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20-00339
Record Dates: First submitted 2020-09-25; First posted 2020-09-29 (Actual); Last update posted 2022-07-22 (Actual); Status verified 2022-07

CONDITIONS: Pulmonary Disease
MeSH Terms: conditions — Lung Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Delayed Lung Transplantation (Experimental): Patients that received lung(s) delayed for transplantation
  Interventions: Procedure: Delayed Lung Transplantation
- Conventional Lung Transplantation (Active Comparator): Reference Therapy
  Interventions: Procedure: Conventional Lung Transplantation

INTERVENTIONS:
Procedure: Delayed Lung Transplantation — Transplants with a planned recipient anesthesia start time between 10:00 pm and 6:00 am will be allowed to move to a start time between 6:00 am and 8:00 am at the earliest. Donor lung(s) cross clamp time must occur between 5:00 pm and 4:00 am. Lungs that meet criteria will be transported in the usual fashion in a cooler of ice at 4oC. Upon arrival to NYULH, the lungs will be transferred to cold static preservation at 10oC within a specific incubator located in a NYULH OR (MYTEMP™65HC, Benchmark Scientific).
  Arms: Delayed Lung Transplantation
Procedure: Conventional Lung Transplantation — Reference Therapy
  Arms: Conventional Lung Transplantation

SUMMARY:
This is a prospective, single-arm study to demonstrate the proof-of-concept of semi-elective lung transplantation. We plan to evaluate 15 patients that receive lung(s) delayed for transplantation under our study criteria.

ELIGIBILITY:
Inclusion Criteria:

* Recipient is ≥ 18 years old
* Recipient, or their Legally Authorized Representative is able and willing to sign informed consent
* Recipient meets standard listing criteria for lung transplantation

Exclusion Criteria:

* Donor lungs meet criteria for transplantation with ex vivo lung perfusion (EVLP)
* Recipient is < 18 years old
* Recipient, or their Legally Authorized Representative is unable to sign informed consent for re-transplantation
* Recipient has any condition that, in the opinion of the Investigator, would make study participation unsafe or would interfere with the objectives of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2020-11-30 (Actual); Primary Completion 2021-12-03 (Actual); Study Completion 2021-12-03 (Actual)

PRIMARY OUTCOMES:
Incidence of ISHLT primary graft dysfunction grade 3 at 72 hours post-transplant | 72 hours
  As defined by International Society of Heart and Lung Transplantation (ISHLT)

CONTACTS AND LOCATIONS:
Overall Officials: Nader Moazami, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset used in the published manuscript will be shared upon reasonable request beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research provided the investigator who proposes to use the data executes a data use agreement with NYU Langone Health. Requests may be directed to the PI. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication
Access Criteria: Requests may be directed to the PI.